CLINICAL TRIAL: NCT00465920
Title: Development and Pilot Evaluation of Modified Cognitive Behavioural Therapy for Adolescents With Early Onset Psychosis
Acronym: mCBT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Collaborators: Goethe University (Other); University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01GV0619
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Psychotic Disorders; Schizophrenia; Schizoaffective Disorder; Delusional Disorder; Schizophreniform Disorder
Keywords: schizophrenia; cognitive behavioural therapy; early onset psychosis; Psychotic disorders (schizophrenia, schizoaffective disorder, delusional disorder, schizophreniform disorder according to DSM IV) in adolescents
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Schizophrenia, Paranoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: modified cognitive behavioural therapy (mCBT)

SUMMARY:
In the last decade cognitive behavioural therapy (CBT) approaches for patients with schizophrenia have been developed, which where especially designed to reduce severity of positive symptoms, readmission rates, treatment non-compliance and disability. Although CBT addresses the key problems of early onset psychoses (EOP)treatment and first evaluations of CBT in adults with schizophrenia are promising, no experience with CBT in adolescents with EOP are available. Therefore the present study is conducted to develop a modified CBT (mCBT) for adolescents with EOP, to explore its acceptance and feasibility and to provide data for a realistic estimation of achievable effect size. Patients are randomized to receive either mCBT+TAU or TAU over a 9 month period. mCBT is an individual outpatient treatment of 20 session and 5 psychoeducational sessions with parents. Follow-ups for two years every 6 months are planned.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia, schizophreniform or schizoaffective disorder (DSM IV 295.1- .9), delusional disorder (DSM IV 297.1)
* Score of 4 or more on one of the PANSS-items P1, P3, G9
* Positive psychotic symptoms for 3 months or more
* Age between 14 and 18
* Fluently German speaking

Exclusion Criteria:

* Diagnosis of delirium, dementia, amnestic or other cognitive disorder, psychiatric disorders due to a somatic factor or related to psychotropic substances according to DSM IV; diseases of the central nervous system
* Alcohol- or drug dependence according to DSM IV
* Verbal IQ < 80
* Travel time to the study centre of more than 1 hour

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-05; Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
PANSS positive syndrome (sum of items P1-P7), assessed during the treatment phase (9 month) monthly and during the follow-up phase (2 years) every 6 months

SECONDARY OUTCOMES:
additional symptom ratings (PSYRATS)
social functioning (GAF)
illness related events (suicide, suicide attempts, rehospitalisation, severe depressive symptom exacerbation)
quality of life (MSLQ)assessed monthly during the treatment phase (9 months) and every 6 months during the follow-up phase (2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bechdolf, PD Dr., Principal Investigator — University of Cologne
Locations (1):
- Department of Psychiatry University Cologne, Cologne, North Rhine-Westphalia, Germany